CLINICAL TRIAL: NCT03681782
Title: Evaluation of the Risks and Benefits of Abdominal Massage Treatment in Neonatalogy in Premature Children
Acronym: PREMASS
Status: Terminated | Type: Observational
Why Stopped: departure of principal investigator with no successor
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 17-015
Record Dates: First submitted 2017-11-16; First posted 2018-09-24 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2022-02

CONDITIONS: Premature Infant
Keywords: premature infant, abdominal massage
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Premature birth creates difficulties for the child in starting his diet and digestion. The immaturity of the major vital functions complicates the abdominal transit. The initial diet, essentially parenteral in the central way, decreases progressively according to the digestive tolerance allowing the increase of the enteral feedings to optimize the growth. To ensure this transition, nurses nurses in Neonatology service, through their knowledge and expertise, practice a daily gesture: abdominal massage-care. This prevents or remedies a slowing of transit. The paramedical clinical examination of the child, determines the realization of this care. Several studies have proved the benefit of massage on the weight gain of premature babies. These stimulate peristalsis, decrease the duration of intestinal transit and the sensations of discomfort and pain related to it. Currently in Neonatology, developmental care (NIDCAP) is an approach to individualized care for the premature to improve its evolution. The fine observation of his behavior allows us to adapt our care and to ensure the respect of his pace. However, the first sensory capacity developed in the fetus, the touch can also be a source of over-stimulation for the premature baby. Moreover, the greater the prematurity, the greater the risk of occurrence of digestive complications. Can the abdominal care-massage in premature babies be harmful or risk increasing existing symptoms? The abdominal care-massage is neither described nor referenced in the nomenclature of nursing, neither taught nor subject to medical prescription.

Few publications exist on this subject, no large-scale research has been reported. On the other hand, the perception of our empirical practice seems to show that the abdominal massage-care is an important aid to the smooth transit of the premature newborn. Transmitted orally by professionals to newcomers to Neonatology, this treatment is carried out in a heterogeneous manner according to professionals. Convinced of its effectiveness, carers wonder about their practice: is there an optimal technique without risk for the child? Determining the absence of risk and the effectiveness of the abdominal care-massage suggests a wider benefit for the well-being and progress of the premature child until he leaves the hospital. This validated practice could be disseminated on a larger scale in other neonatal departments.

ELIGIBILITY:
Inclusion Criteria:

* Children born before 37 weeks of amenorrhea hospitalized in the neonatology department

Exclusion Criteria:

* children with a malformation or a digestive pathology with or without surgery
* medical prescription of non-massage care
* children born under the secret

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children born before 37 weeks of amenorrhea hospitalized
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Change in the neonatal infant pain score | up to 30 days from baseline
  neonatal infant pain scale (EDIN)) (>4 or>=4)
bradycardia | up to 30 days from baseline
  bradycardia (yes/no)
arterail oxygenation desaturation | up to 30 days from baseline
  arterail oxygenation desaturation (yes/no)
Change in the abdominal aspect | up to 30 days from baseline
  bloating, visibility of the abdominal loops, collateral circulation, abdominal staining
Significant adverse effects | up to 30 days from baseline
  volvulus of the small intestine, intestinal perforation

CONTACTS AND LOCATIONS:
Overall Officials: Virginie DELVAL, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided
Publication